CLINICAL TRIAL: NCT06592807
Title: The Effect of Perioperative Warm Socks on Maintaining Body Temperature in Patients Undergoing Spinal Surgery: Randomized Controlled Trial
Brief Title: The Effect of Perioperative Warm Socks on Maintaining Body Temperature in Patients Undergoing Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hatice Merve Alptekin, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023/262
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Spinal Surgery
Keywords: body temperature; perioperative; warm sock; hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers who collected data and analyzed the study results were different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm Sock Group (Experimental): 1. Before surgery, patients are informed about the study and their tympanic body temperatures are measured.
  2. The socks that the patient will wear during the surgery are warmed and put on.
  3. During the surgery, the operating room temperature is measured and recorded. The patient's tympanic body temperature is also measured and recorded. (Every half hour).
  4. When the patient is taken to the postoperative care unit, the socks are changed to new heated socks.
  5. After the surgery, patients are given a survey question regarding socio-demographic data. Patients' pain is assessed with VAS (visual analog scale). Patients' thermal comfort is assessed. Patients' shivering is assessed according to the shivering scale. In addition, patients' vital signs are assessed every 15 minutes for one hour.
  Interventions: Other: Perioperative Warm Socks
- Control Group (No Intervention): 1. Before surgery, patients are informed about the study and their tympanic body temperatures are measured.
  2. During the surgery, the operating room temperature is measured and recorded. The patient's tympanic body temperature is also measured and recorded. (Every half hour).
  3. After the surgery, patients are given a survey question regarding socio-demographic data. Patients' pain is assessed with VAS (visual analog scale). Patients' thermal comfort is assessed. Patients' shivering is assessed according to the shivering scale. In addition, patients' vital signs are assessed every 15 minutes for one hour.

INTERVENTIONS:
Other: Perioperative Warm Socks — The socks to be used in the study were provided by the researcher. The socks were suitable for foot sizes 36-45. The socks were white and made of cotton fabric. The socks were sterilized in an autoclave before use. The socks were put on the patients just before the surgery. The socks were heated to 40 degrees with an intravenous fluid warming machine.The socks remained on the patients feet throughout the surgery. After the surgery, the patients socks were removed and new heated socks were put on. The socks were kept on the patients feet for 1 hour. All socks were used for single use.
  Arms: Warm Sock Group

SUMMARY:
It is important to maintain the body temperature of patients during spine surgery because hypothermia that occurs during surgery can increase the risk of complications and negatively affect the recovery process. For this reason, various methods are being investigated to maintain the body temperature of patients during and after surgery. Warm socks application is a simple and effective method performed by putting warm socks on the feet of patients. This application has been shown to better maintain the body temperature of patients during the perioperative period and may reduce the incidence of hypothermia. Warm socks help maintain body temperature by increasing blood circulation and reducing heat loss. As a result, warm socking application is considered a useful and recommended method for maintaining body temperature in patients undergoing surgery.

DETAILED DESCRIPTION:
Hypothermia during surgery is a common problem among patients undergoing surgery. It is known that approximately half of the patients who undergo surgery develop hypothermia. Hypothermia is defined as a central temperature below 36°C. The body temperature of patients decreases during the first hour of general anesthesia and continues to decrease when the surgery exceeds 2 hours. In the event of hypothermia, the patient develops a physiological shivering response. It can also increase patients oxygen consumption by up to 40%. Active and passive heating methods are used to prevent this. Warm socks are one of the passive heating methods.

In the preoperative period, putting pre-warmed socks on patients is effective in maintaining core body temperature, controlling shivering response and ensuring thermal comfort of patients. Pre-warmed socks are a noninvasive, easy-to-wear, painless and cost-effective method to prevent body temperature loss. The application of warm socks is also a method that allows the patient position to be changed and surgical preparation, is comfortable for the patient, reduces preoperative anxiety and can be applied without a physician order.

Study Population and Sampling: The universe of the study will consist of patients who underwent spinal surgery in the Operating Room of Istanbul Bakırköy Prof. Dr. Mazhar Osman Mental Health and Nervous Diseases Education and Research Hospital on the specified dates.

Sample: In the study, Gpower was used to determine the effect of perioperative warm socks application on maintaining body temperature in patients undergoing spinal surgery. The study findings reported by Lee et al. were used to determine the d value, which is the effect size index. It was calculated as α= 0.05, power=0.80 d=0.63. The sample was determined as 32 people for each group, a total of 64 patients.

Randomization: The research was conducted as double blind randomized and controlled experimental study. A simple computer-assisted randomization method was used to distribute the groups homogeneously.

For this purpose, 64 sets were created by using the functions on the internet address ;https://www.random.org/integer-sets; and each of these sets included 8 subjects, 4 subjects from each study group. As the next process, 64 sets were shown with 1 number each, 8 numbers between 1 and 64 were generated using the ;RANDOMLY SEARCH; function in Excel, and 8 sets to be used in randomization were randomly determined. Each set will contain 8 (4 experimental, 4 control) patients.

Data Collection Method: Data were collected by the researcher using face-to-face interview technique.

Data Collection Tools:

Personal information form (sociodemographic characteristics): This form, prepared by the researcher in line with the literature, aims to obtain information about the participants; sociodemographic characteristics (gender, age, occupation, etc.) and the surgery (duration of the surgery, start and end time of the surgery, etc.).

Tympanic temperature table: It was measured just before the surgery and continued to be measured every half hour throughout the surgery.

Operating room temperature table: It was measured just before the surgery and continued to be measured every half hour throughout the surgery.

Shivering scale: To determine the degree of the patients shiver, the researcher observed the patient. Then, patient gave a score between 0 and 4 to rate. 0: No signs of shiver. 4: Mean teeth chattering shiver. Measured after surgery.

Subjectıve thermal comfort scale: The patient was asked to determine the temperature he felt. It was evaluated between 1 and 6. 1: very cold, 6: very hot. It was measured after the surgery.

Vital signs: Body temperature, pulse, respiration, blood pressure, and SpO2 values were measured every 15 minutes for the first hour after surgery.

Visual analog scale: The two extreme definitions of the parameter to be evaluated are written at both ends of a 100 mm line, and the patient is asked to indicate where his/her own condition fits on this line by drawing a line, putting a dot, or marking. For example, for pain, I have no pain at one end, and very severe pain is written at the other end, and the patient marks his/her current condition on this line. The length of the distance from the place where there is no pain to the point marked by the patient indicates the patients pain.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 18-64 years old
* Able to understand and speak Turkish
* In the ASA1,2,3 class according to the ASA classification
* Not have anemia, coagulation problems, peripheral circulation disorders or a metabolic disease
* Willing to undergo spine surgery (LDH,SDH, scoliosis, stabilization)
* Not undergoing spinal and local anesthesia
* Volunteering to participate in the study

Exclusion Criteria:

* The patient's surgery lasting less than 2 hours or more than 5 hours
* The patient's socks are removed during the surgery
* The patient's tympanic body temperature is not checked during the surgery
* Complications develop during and after the surgery
* The patient is taken to intensive care immediately after the surgery

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
Tympanic temperature measurement | Every half hour during the surgery. (Until the 5th hour)
  It is the measurement of the patient's temperature via the tympanic route.
Shivering | It measured once at the 1st minute after surgery.
  To determine the degree of the patient shiver, the researcher observed the patient. Then, patient gave a score between 0 and 4 to rate. 0: No signs of shiver. 4: Mean teeth chattering shiver.

SECONDARY OUTCOMES:
Subjectıve thermal comfort | It measured at the 15th minutes after surgery.
  The patients were asked to determine the temperature they felt. It was evaluated between 1 and 6. 1: very cold, 6: very hot.
Visual analog scale: Pain | It measured at the 15th minutes after surgery.
  The two extreme definitions of the parameter to be evaluated are written at both ends of a 100 mm line, and the patient is asked to indicate where his/her own condition fits on this line by drawing a line, putting a dot, or marking. For example, for pain, I have no pain at one end, and very severe pain is written at the other end, and the patient marks his/her current condition on this line. The length of the distance from the place where there is no pain to the point marked by the patient indicates the patients pain.
Body temperature | Measured every 15 minutes for the first hour after surgery.
  It is the measurement of the patients temperature via the tympanic route
Pulse | Measured every 15 minutes for the first hour after surgery.
  Measurements were made from the patients index finger with a pulse oximeter.
Spo2 | Measured every 15 minutes for the first hour after surgery.
  Measurements were made from the patients index finger with a pulse oximeter.
Respiration | Measured every 15 minutes for the first hour after surgery
  The patients breathing was counted for 1 minute.
Blood pressure | Measured every 15 minutes for the first hour after surgery.
  The patient was monitored by placing a cuff on patients arm to measure his blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Merve Alptekin, PhD, Principal Investigator — Kocaeli University
Locations (1):
- Hatice Merve Alptekin, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Frisch NB, Pepper AM, Rooney E, Silverton C. Intraoperative Hypothermia in Total Hip and Knee Arthroplasty. Orthopedics. 2017 Jan 1;40(1):56-63. doi: 10.3928/01477447-20161017-04. Epub 2016 Oct 27. PMID 27783839
- [Background] Kim, J. S. (2004). Anesthesia and body temperature. Korean Journal of Anesthesiology, 47(5), 609-616.
- [Background] Collins, V. J. (1996). Temperature regulation and heat problems. In V. J. Collins (Ed.), Physiologic and pharmacologic bases of anesthesia (pp. 316-344). Baltimore, MD: Williams & Wilkins.
- [Background] Shakya S, Chaturvedi A, Sah BP. Prophylactic low dose ketamine and ondansetron for prevention of shivering during spinal anaesthesia. J Anaesthesiol Clin Pharmacol. 2010 Oct;26(4):465-9. PMID 21547171
- [Background] Lee HY, Kim G, Shin Y. Effects of perioperative warm socks-wearing in maintaining core body temperature of patients undergoing spinal surgery. J Clin Nurs. 2018 Apr;27(7-8):1399-1407. doi: 10.1111/jocn.14284. Epub 2018 Mar 26. PMID 29396880
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665